CLINICAL TRIAL: NCT02903862
Title: Caregivers Virtual Health eBrain Study II
Brief Title: Health-eBrain Study
Acronym: HeB
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not meet enrollment requirement.
Sponsor: AnthroTronix, Inc. (Industry)
Collaborators: Bright Focus Foundation (Unknown); Mindoula Health Inc. (Unknown); 21st Century Brain Trust (Other); Geoffrey Beene Foundation (Unknown)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 091614A
Record Dates: First submitted 2016-08-03; First posted 2016-09-16 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Depression and Burden in Caregivers
Keywords: Caregivers; Case Management; Alzheimer's Disease; Cognition; Caregiver Burden; Depression
MeSH Terms: conditions — Depression; Alzheimer Disease; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Arm (Experimental): Participants will receive the intervention, Mindoula plus DANA, which involves working with a case manager via an app for 12 weeks. The case manager will help the participant cope with the stresses of caregiving as well as remind them to use the DANA cognitive assessment app. This arm will also take the study's psychological surveys.
  Interventions: Behavioral: Mindoula; Device: DANA
- Waitlist Control Arm (Other): These participants will take psychological surveys and a usability questionnaire for the first 12 weeks of participation, then, for the 12 weeks following, take the psychological surveys along with DANA and a usability questionnaire.
  Interventions: Device: DANA

INTERVENTIONS:
Behavioral: Mindoula — The Mindoula intervention is a combination of case management and a messenger application. Case managers monitor how the participant is doing and any needs and provide 24/7 support & assistance, including care coordination, treatment adherence, and matching the participant with providers and community resources. Each participant will be given an intake questionnaire to establish goals and behavioral health history. Participants will use the app and work with the case manager for 12 weeks.
  Arms: Intervention Arm
Device: DANA — DANA is an FDA-cleared neurocognitive assessment software administered on a smartphone or tablet to measure changes in cognitive efficiency. DANA also includes Ecological Momentary Assessments to track mood, sleep, stress, and memory. Intervention participants will take DANA weekly. The Waitlist Control arm will take DANA weekly 12 weeks after enrollment.

SUMMARY:
The purposes of this study are to (1) track dementia caregiver health indicators over 12 weeks, both with and without the Mindoula plus DANA intervention (case manager and mobile messaging and assessment applications) to determine if the intervention improves caregiver health and (2) obtain feedback from caregivers to inform on the design of future interventions.

DETAILED DESCRIPTION:
This study will track the mental status and cognition of caregivers with and without the Mindoula and DANA intervention and use subject feedback to aid in designing future interventions for caregivers.

This is a remotely administered, virtual study targeting dementia caregivers who are mild to moderately depressed. Screening calls for online administration of four surveys to determine inclusion in the study arms. These surveys will be taken on the Health-eBrain website, both at baseline/screening and throughout participation. All other participation will be completed on the participant's mobile phone, and all psychological and cognitive tests will be self-administered.

This study has a between-group design. Participants will be screened for eligibility and then randomized into each arm. The intervention arm will receive the Mindoula plus DANA intervention. The wait list control arm will take the psychological surveys at regular intervals then, after 12 weeks, be enrolled in the DANA-only observation group. The DANA-only group will take DANA and a usability questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Females and males who regularly provide care for a person with Alzheimer's Disease
* Between the ages of 45-75
* Self-reported ability to speak and read English
* Providing care for at least a year

Participants in the Intervention and Waitlist Control Arms must meet the following additional inclusion criteria:

* Zarit Burden Inventory (ZBI) Score of 9+
* Overall M3 score of 33+
* M3 Depression score of 7+
* Female Only
* Minimum hours of caregiving a week must be equal to or greater than 20 hours

Exclusion Criteria:

* Anyone with a known cognitive diagnosis
* Anyone with color blindness
* Overall score of high risk on the M3 and/or high risk on the PTSD or Bipolar subsection of the M3
* Failure to meet all inclusion criteria per arm

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline M3 Behavioral Scale score over 12 weeks | At baseline, and 4, 8, and 12 weeks.

SECONDARY OUTCOMES:
Change from baseline Zarit Burden Inventory score over 12 weeks | At baseline, and 4, 8, and 12 weeks.
Change from baseline PROMIS Sleep Disturbance Short Form 8a score over 12 weeks | At baseline, and 4, 8, and 12 weeks.

OTHER OUTCOMES:
Usability Questionnaire | At baseline, and 4, 8, and 12 weeks.
  Survey on using DANA that will help the researchers better understand the development of technologies for this population
Paired Associates Learning | At baseline and 12 weeks
  The PAL assesses visual memory and new learning.
PERMA Profiler | At baseline and 12 weeks
  This survey assesses five core element of psychological well-being and happiness - Positive emotions, Engagement, Relationships, Meaning, and Accomplishments - as well as subjective wellbeing and sense of loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Corinna E Lathan, Ph.D, Principal Investigator — AnthroTronix, Inc.
Locations (1):
- AnthroTronix Inc, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lathan C, Wallace AS, Shewbridge R, Ng N, Morrison G, Resnick HE. Cognitive Health Assessment and Establishment of a Virtual Cohort of Dementia Caregivers. Dement Geriatr Cogn Dis Extra. 2016 Mar 22;6(1):98-107. doi: 10.1159/000444390. eCollection 2016 Jan-Apr. PMID 27099613
- See also: Website where study is being conducted. Participants register and take their psychological surveys here. — http://www.health-ebrainstudy.org